CLINICAL TRIAL: NCT05429645
Title: Cardiac Resynchronization Under Electroanatomical Guidance After Failure of Primary Implantation: CRT3D Study
Brief Title: Cardiac Resynchronization Under Electroanatomical Guidance After Failure of Primary Implantation
Acronym: CRT3D
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A new technique has rendered the study technique obsolete, making it inappropriate to continue the study due to lack of therapeutic interest.
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A00811-42
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Anomaly
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3-dimensional guidance technique (Experimental): 3-dimensional (3D) guidance technique to position the heart probes in the setting up of a pace maker
  Interventions: Procedure: setting up of the pace maker

INTERVENTIONS:
Procedure: setting up of the pace maker — Setting up of a pace maker using a 3-dimensional (3D) guidance technique

SUMMARY:
The purpose of the study is to assess the feasibility of cardiac resynchronization under electroanatomic guidance in the event of primary implantation failure due to catheterization failure or instability in the coronary sinus ostium

DETAILED DESCRIPTION:
As part of this study, to avoid surgery, the doctor will use a 3-dimensional (3D) guidance technique to position the heart probes in an optimal position during a new endovascular intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient with indication for implantation of a classic multisite pacemaker;
* New York Heart Association II/IV patient despite optimal medical treatment;
* Patient with left ventricular ejection fraction ≤35%;
* Patient with a widened QRS > 120ms;
* Patient with at least one lateral coronary sinus vein visualized on angiography during the 1st procedure (if performed);
* Patient with failure of resynchronization via the endovenous route due to difficulty in accessing the coronary sinus or instability in the coronary sinus;
* Patient having been informed and having signed an informed consent form;
* Patient able to understand the information related to the study (absence of linguistic, psychological, cognitive problem, etc.), and to complete questionnaires.

Exclusion Criteria:

* Patient with resynchronization failure due to occlusion of the superior vena cava;
* Patient with no usable lateral coronary sinus vein;
* Patient with a life expectancy < 3 months;
* Patient wearing a vena cava filter;
* Patient with active sepsis;
* Pregnant or likely to be pregnant (of childbearing age, without effective contraception) or breastfeeding;
* Patient participating in another clinical trial, or in a period of exclusion from another clinical trial;
* Patient not benefiting from a social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Setting up with success of the Left Ventricular lead | during the time of the setting up of the pace maker
  Feasibility of cardiac resynchronization under 3 dimension assistance in the event of primary implantation failure will be assessed by the proportion of patients for whom the Left Ventricular lead has been placed successfully with a pacemaker

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Le Bois, Lille, France

IPD SHARING:
Plan to Share IPD: No